CLINICAL TRIAL: NCT06269965
Title: Assessment of Collagen Membrane Interest in Distal Cuff Lesions Repair
Acronym: REGENECUFF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-A02181-44
Record Dates: First submitted 2024-02-13; First posted 2024-02-21 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Cuff Rotator Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regeneten® Arm (Experimental): Arthroscopic shoulder repair, in double row, with complete coverage of the foot print and addition of Regeneten®
  Interventions: Device: Regeneten® adding
- Witness Arm (No Intervention): Arthroscopic shoulder repair, in double row, with complete coverage of the foot print

INTERVENTIONS:
Device: Regeneten® adding — Arthroscopic shoulder repair, in double row, with complete coverage of the foot print and addition of Regeneten®
  Arms: Regeneten® Arm

SUMMARY:
Rotator cuff refers to a set of 4 shoulder tendons. These tendons are the sub-scapularis, supra-spinatus, infra-spinatus and teres minor. Rotator cuff tear corresponds to total or partial tendon disinsertion at the greater tuberosity level or a few centimeters in upstream.

Rotator cuff surgery is an increasingly popular procedure practiced in France. In limited cuff lesions (distal or intermediates) and in absence of contraindication, absence of tendons' healing is around 10 to 20%. Sofcot estimates that 90% of caps' heals remain healed 10 years after surgery in distal lesions. However, even in case of a healed cuff, if tendon quality is not good, function will be impaired.

Bioinductive implant Regeneten® is an advanced healing solution for biological improvement and regeneration of tendons on all types rotator cuff tear. A randomized study was initiated whose main objective was to evaluate integrity of repaired tendon with MRI one year after intervention according to Sugaya's classification. Results showed a recurrence rate of 8.3% in Regeneten® group compared to 25.8% in witness group.

In this context, this study is based on hypothesis that adding Regeneten® during rotator cuff repair could be beneficial on tendon healing rate but also on tendon quality healing.

DETAILED DESCRIPTION:
Rotator cuff refers to a set of 4 shoulder tendons. These tendons are the sub-scapularis, supra-spinatus, infra-spinatus and teres minor. They are located at the head of arm bone (humerus) and cover it, hence the name "cap".

Shoulder tendon injuries occur following sport's trauma, microtraumas often falling within the framework of musculoskeletal disorders (MSD) and heavy professional practices, or they are more simply due to body natural aging.

Rotator cuff tear corresponds to total or partial tendon disinsertion at the greater tuberosity level (part of humerus where the supraspinatus and infraspinatus tendons insert) or a few centimeters in upstream. This disinsertion creates a passage between glenohumeral joint and subacromial space. Subsequently, rupture can extend forwards or backwards (which is the most common frequent case).

Rotator cuff surgery is an increasingly popular procedure practiced in France. Regardless of technical progress allowing today an ambulatory arthroscopic surgery, its success comes also from better knowledge of its indications and its clinical and histological results.

Overall, in limited cuff lesions (distal or intermediates) and in absence of contraindication, absence of tendons' healing is around 10 to 20%. Sofcot estimates that 90% of caps' heals remain healed 10 years after surgery in distal lesions. However, even in case of a healed cuff, if tendon quality is not good, function will be impaired. Bioinductive implant Regeneten® is an advanced healing solution for biological improvement and regeneration of tendons on all types rotator cuff tear. A randomized study (NCT04444076) was initiated whose main objective was to evaluate integrity of repaired tendon with MRI one year after intervention according to Sugaya's classification. Results showed at one year follow-up a recurrence rate of 8.3% in Regeneten® group compared to 25.8% in witness group.

In this context, this study is based on hypothesis that adding Regeneten® during rotator cuff repair could be beneficial on tendon healing rate but also on tendon quality healing.

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, aged ≥ 18 years
* Patient candidate for rotator cuff repair affecting supraspinatus tendon (distal lesion) +/- infraspinatus on a non-pseudo-paralytic shoulder +/- proximal lesion of subscapularis
* Patient with GI ≤ 2 for each muscle
* Non-smoking patient
* Patient who is not involved in a work accident
* Patient candidate for total rotator cuff repair completely covering the footprint during surgery

Exclusion Criteria:

* Patient with contraindication to MRI
* Patient operated for cuff revision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2024-03-15 (Estimated); Primary Completion 2027-04-15 (Estimated); Study Completion 2027-04-15 (Estimated)

PRIMARY OUTCOMES:
Rotator cuff healing quality | Year one
  Rotator cuff healing quality is evaluated with classification of Sugaya varying from type I to type V (performed from MRI) :
  type I: sufficient thickness compared to normal cuff with homogeneous low signal
  type II: sufficient thickness compared to normal cuff with partial high-intensity area
  type III : <50% thickness compared to normal cuff without discontinuity suggests partial-thickness delamination tear
  type IV : minor discontinuity (1-2 slices) on both oblique coronal and oblique sagittal images suggests small full-thickness tear
  type V : major discontinuity (>2 slices) on both oblique coronal and sagittal images suggests medium or large full-thickness tear

IPD SHARING:
Plan to Share IPD: No